CLINICAL TRIAL: NCT00066391
Title: Phase II Study of Irinotecan (CPT 11) and Cisplatin (CDDP) in Metastatic or Locally Advanced Penile Carcinoma
Brief Title: Irinotecan and Cisplatin in Treating Patients With Locally Advanced or Metastatic Penile Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: EORTC-30992; EORTC-30992
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Penile Cancer
Keywords: penile squamous cell carcinoma; stage III penile cancer; stage IV penile cancer
MeSH Terms: conditions — Penile Neoplasms | interventions — Cisplatin; Irinotecan; Neoadjuvant Therapy

INTERVENTIONS:
Drug: cisplatin
Drug: irinotecan hydrochloride
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as irinotecan and cisplatin use different ways to stop tumor cells from dividing so they stop growing or die. Combining irinotecan with cisplatin may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining irinotecan with cisplatin in treating patients who have locally advanced or metastatic penile cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the anticancer activity of irinotecan and cisplatin in patients with locally advanced or metastatic penile cancer.
* Determine the objective response rate and duration of response in patients treated with this regimen.
* Determine the acute side effects of this regimen in these patients.

OUTLINE: This is an open-label, nonrandomized, multicenter study.

Patients receive irinotecan IV over 30 minutes on days 1, 8, and 15 and cisplatin IV over 1-3 hours on day 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients not undergoing local treatment receive up to 8 courses. Patients planning to undergo surgery receive up to 4 courses.

Patients are followed every 8 weeks until disease progression and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 13-28 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed penile squamous cell carcinoma

  * Locally advanced or metastatic disease

    * T3, N1-2 OR T4, N3, M1
* Measurable disease outside of any previously irradiated field
* No clinical signs of brain metastases

PATIENT CHARACTERISTICS:

Age

* 75 and under

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN (5 times ULN in the presence of liver metastases)
* Transaminases no greater than 2.5 times ULN (5 times ULN in the presence of liver metastases)

Renal

* Glomerular filtration rate at least 60 mL/min

Gastrointestinal

* No chronic diarrhea
* No unresolved bowel obstruction
* No chronic inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis)

Other

* No other prior or concurrent malignancy except adequately treated skin cancer
* No psychological, familial, sociological, or geographical condition that would preclude study compliance and follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy
* No concurrent radiotherapy for pain control

Surgery

* Not specified

Other

* No other concurrent experimental or anticancer therapy

Max Age: 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-06; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Objective response rate measured by RECIST at 8 weeks after completion of study treatment

SECONDARY OUTCOMES:
Duration of response as measured by Kaplan-Meier every 8 weeks until progression, and then every 3 months thereafter
Toxicity as measured by NCI-CTC v2.0 every 8 weeks until progression

CONTACTS AND LOCATIONS:
Overall Officials: Christine Theodore, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (8):
- U.Z. Gasthuisberg, Leuven, Belgium
- Institut Gustave Roussy, Villejuif, France
- National Institute of Oncology, Budapest, Hungary
- Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam, Netherlands
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland
- United Kingdom (3):
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Saint Bartholomew's Hospital, London, England

REFERENCES:
- [Result] Theodore C, Skoneczna I, Bodrogi I, Leahy M, Kerst JM, Collette L, Ven K, Marreaud S, Oliver RDT; EORTC Genito-Urinary Tract Cancer Group. A phase II multicentre study of irinotecan (CPT 11) in combination with cisplatin (CDDP) in metastatic or locally advanced penile carcinoma (EORTC PROTOCOL 30992). Ann Oncol. 2008 Jul;19(7):1304-1307. doi: 10.1093/annonc/mdn149. Epub 2008 Apr 15. PMID 18417462